Version Date: 27 February 2023

Treating Loneliness in Students: a Pilot Trial on the Feasibility and Acceptability of a Value-Based Social Approach Cognitive Behavioural Intervention

**Central Contact Person** 

Carmen van den Bulck, MSc Telephone: +31634570181

Email: <u>c.m.m.vandenbulck@uva.nl</u>

University of Amsterdam

#### TITLE OF THE STUDY: LET'S GET SOCIAL

Dear participant,

Welcome to the course and study "Let's get Social", of the Faculty of Social and Behavioural Sciences of the University of Amsterdam (UvA).

It is important that you learn about the procedure of this course and the accompanying study before it starts, so please read the following text carefully. If anything is unclear to you, feel free to ask the researcher directly, or contact them through email: <a href="mailto:c.m.m.vandenbulck@uva.nl">c.m.m.vandenbulck@uva.nl</a>. The researcher will be happy to answer any questions you may have.

#### Goal of the course and study

Loneliness is, in principle, a healthy emotion that can affect anyone. When you feel lonely, this is a signal that motivates you to reconnect with other people. Negative emotions and thoughts can hinder this, making it difficult to (re)connect with others. In that case, loneliness can become chronic. In the course "Let's get Social", you will train skills that help reducing feelings of loneliness and increase social connection. The accompanying study evaluates the effects of this course.

#### The course

During the course, you will learn various skills that can help you to alleviate loneliness by (re)connecting with others. The sessions will be given in small groups of around seven students and two trainers. The trainers are employees of the UvA Clinical Psychology department. Each session will give some background information on a particular aspect of loneliness. We will then use exercises focusing on this aspect and you will learn skills that that you can use to address these issues. We will practice these skills during the session, but you will also continue to practice them in your daily life in between the sessions.

Participating in the course will probably require a change in your social behaviour and this may feel new or even uncomfortable in the beginning. Training new skills takes effort and the tension involved is normal. As you will practice with these situations, it is expected that you will benefit from it in the end. It is important that there is a safe environment for participants. During the course, there is room to tell personal things and be open about why you find certain exercises difficult. Both the trainers and the participants will treat this confidentially.

#### Procedure of the course and study

The course consists of seven weekly 2-hour sessions and one booster session and starts in May 2023. In the week of March 13, a screening will be planned to see whether the course is suitable for you. This involves answering several online questionnaires an a Zoom interview with one of the trainers to assess various psychological symptoms. The screening procedure takes approximately 45 minutes. If you are eligible, you will be invited to participate in the study.

As we want to study the effects of the course, we will ask you to complete several questionnaires before, during, and after the course. These questionnaires are about your mood, anxiety, and level of loneliness. During the 7-week period leading up to the course, you will receive short weekly questionnaires that take 1-2 minutes to complete. After a pre-test (10 minutes), the course begins in May and you will continue to complete short weekly questionnaires throughout the course. Finally, you will complete a post-test (10 minutes) as well as a one-month follow-up (10 minutes) and a three-month follow-up (10 minutes) after the course ends. The answers you give to all these questionnaires will remain confidential and will be processed anonymously.

Audio recordings will be made of all group sessions. We do this to monitor and improve the quality of the course. The UvA researchers involved in this study will listen to the recordings to carry out quality checks. Only the researchers involved in this study will have access to the audio recordings.

#### Voluntary participation

Your participation in this study is voluntary: you are not obligated to participate. You may decide to stop your participation during the study, and you can also decide to withdraw after the study. You do not have to provide a reason for stopping. If you decide to stop, your (personal) data will be deleted upon request, except for (personal) data that have already been processed. There are no consequences to stopping. You can indicate directly to the researcher that you wish to withdraw from participation, or you can contact the following email address: <a href="mailto:c.m.m.vandenbulck@uva.nl">c.m.m.vandenbulck@uva.nl</a>. Additionally, because this study can be emotionally taxing, the Ethics Review Board of the Faculty of Social and Behavioral Sciences allows you to request the researcher to remove your (personal) data within two days. If you wish to do so, contact the researcher through this email address: <a href="mailto:c.m.m.vandenbulck@uva.nl">c.m.m.vandenbulck@uva.nl</a>

#### **Privacy**

We treat your personal data confidentially, as required by law (the General Data Protection Regulation or GDPR). Personal data are data that can be traced back to you individually, either directly or indirectly. When working with (personal) data, researchers may use external parties, for instance when administering online surveys. In that case the appropriate contracts with these parties have been arranged in order to warrant your privacy.

#### **Collaborations**

In this study your research data are processed only by UvA researchers.

#### Data sharing

The results of this study may be shared with other researchers and/or may be shared through a public database (open access), without any (directly identifying) personal data. Non-identifiable data may be used in other future research, which may investigate a different topic than the study you are currently participating in.

Version Date: 27 February 2023

#### Retention period

Research data, including personal data that are needed to answer the research question, will be retained for at least 10 years. Your contact details will be deleted as soon as possible.

#### **Further information**

If you have any questions about the study, either before you participate or afterwards, please feel free to contact the responsible researcher: Carmen van den Bulck (c.m.m.vandenbulck@uva.nl). You can direct any formal complaints about this study to the member of the Ethics Review Board of the Faculty of Social and Behavioral Sciences of the University of Amsterdam, Wery van den Wildenberg (W.P.M.vandenWildenberg@uva.nl). If you have any questions or complaints about the processing of your personal data, you can also contact the Data Protection Officer of the University of Amsterdam through fg@uva.nl.

With kind regards,

Carmen van den Bulck, MSc

Email: <u>c.m.m.vandenbulck@uva.nl</u>

# DECLARATION OF CONSENT \*Offline research\*

This form supplements the written information you have received about the study in which you are participating. If you sign this form, you declare that you have read and understood the information, and that you agree to the procedure as described in the information letter.

For further information about this study, please contact the responsible researcher, Carmen van den Bulck (c.m.m.vandenbulck@uva.nl). Should you have any complaints about this study, please direct them at the member of the Ethics Review Board, Tinka Beemsterboer (datasteward-psy@uva.nl). If you have any questions or complaints about the processing of your personal data, you can also contact the Data Protection Officer of the University of Amsterdam through fg@uva.nl.

## Signed in duplicate

# [PARTICIPANT]

- I am 16 years or over.
- I have read and understood the provided information.
- I agree to participate in this study, and I consent to the use of the resulting data.
- I maintain the right to revoke this consent without giving any reason.
- Name of participant

  Signature of participant

  Signature of participant

  Date

## [RESEARCHER]

| <ul> <li>I have informed the participant about the study.</li> <li>I am willing to answer any questions that may still arise to the best of my abilities.</li> </ul> | |
|---|---|
| Name of researcher | Signature of researcher |
| Date | |